CLINICAL TRIAL: NCT01434043
Title: Diagnostic Accuracy of Cardiac CT Perfusion Compared to PET Imaging
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Kelley Branch, Associate Professor, Medicine/Cardiology, University of Washington
Other Study IDs: STUDY00001616
Record Dates: First submitted 2011-09-09; First posted 2011-09-14 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Myocardial Ischemia; Coronary Artery Disease; Myocardial Infarction
Keywords: Cardiac CT perfusion; Positron emission tomography perfusion; Quantitative perfusion
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Myocardial ischemia patients

SUMMARY:
This purpose of this research project is to test the diagnostic accuracy (i.e., sensitivity, specificity, positive and negative predictive value, and receiver operator curve area under the curve) of cardiac computed tomography (CT) perfusion as compared to the best non-invasive test of blood flow -- cardiac positron emission transmission (PET) perfusion imaging.

The primary outcome of the study is to determine the CT perfusion technique with the highest overall diagnostic accuracy measured by the highest area under the receiver operator curve.

The investigators will test 4 different CT perfusion techniques. (A) Qualitative, visual inspection of the contrast-enhanced CT images (B) Enhanced voxel distribution analysis (C) Rate of myocardial contrast enhancement analysis (D) Quantitative heart blood flow using a distributed 2-region analysis

A second aim is to reduce the radiation dose needed to maintain CT perfusion diagnostic accuracy. Using the CT perfusion data, the investigators will model the minimal number of cardiac cycle radiation exposures needed to keep the diagnostic accuracy similar to the full data set.

A third aim is to test the incremental diagnostic accuracy of CT angiography plus CT perfusion to identify regions of low blood flow as compared to PET perfusion alone.

DETAILED DESCRIPTION:
Chest pain and other symptoms can occur as a result of blockages in the arteries that supply the heart; these arteries are called the "coronary arteries". Blockages in the coronary arteries may decrease blood flow and oxygen delivery to the heart muscle, causing chest pain or other "anginal" symptoms. Coronary angiography is a commonly used test to visualize coronary artery disease or blockages but may not provide all the answers physicians need to assess patients with symptoms like chest pain. Two options for coronary angiography exist, invasive angiography and cardiac computed tomography angiography (CCTA). CCTA is completed by injecting contrast into a peripheral vein (not an artery) and then imaging when the coronary arteries fill with contrast. The imaged coronary arteries may be blocked partially, completely or not at all. While a blockage that occludes greater than 70% of an artery is highly correlated with chest pain or other anginal symptoms, occlusions of 40% or more may or may not decrease heart blood flow. Often multiple imaging studies are needed to evaluate whether blood flow is decreased in the setting of partial coronary artery blockages including non-invasive heart imaging to assess heart blood flow.

One type of nuclear imaging is termed positron emission tomography (PET). In order to differentiate blockages that have poor heart perfusion with activity, nuclear PET images are taken at rest, when flow should be normal, and then repeated after the investigators "stress" the heart with medications. If blood flow is decreased during stress, a "defect" on the PET images is seen.

An alternative, non-invasive technique to test for heart blood flow/perfusion to to measure heart blood flow as computed tomography (CT) contrast goes in and comes out. Preliminary studies in animals and humans to assess heart blood flow/perfusion using contrast-enhanced cardiac CT have been promising, but further work is needed. Combining CCTA with CT blood flow/perfusion measurements in the same setting could lead to a single, accurate diagnostic test that measures coronary artery blockage as well as blood flow.

One limitation of CT imaging is the amount of radiation that can be given. The CCTA radiation dose is currently less than both nuclear PET imaging and invasive coronary angiography. However, if CT blood flow imaging is added to routine CCTA to assess heart perfusion and coronary blockages in one test, the radiation dose may be higher.

The primary purpose of this research project is to test the diagnostic accuracy of various cardiac CT perfusion techniques as compared to the best non-invasive test of blood flow, cardiac PET perfusion imaging. The investigators goal is to use the least amount of radiation to achieve a high diagnostic accuracy for CCTA as well as CT blood flow/perfusion. The investigators goal is to have CT heart blood flow/perfusion radiation doses that are the same or less than nuclear blood flow imaging. The investigators have estimated that they need as few as 4 low radiation dose images of the heart to allow accurate heart blood flow measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for

  1. clinically indicated PET imaging for assessment of myocardial ischemia
  2. clinically indicated CCTA scanning with known coronary artery disease
* ≥20 years of age and ≤ 80 years of age
* Able to provide written informed consent

Exclusion Criteria:

* Contraindications to beta blockers or regadenoson

  * Active reactive airway disease
  * 2nd or 3rd degree heart block (without a pacemaker)
  * Sick sinus syndrome (without a pacemaker)
  * Long QT syndrome (QTC > 500 msec)
  * Severe hypotension
  * Decompensated heart failure
* Pregnancy
* Contraindications to undergoing any CT imaging procedure with contrast:

  * Irregular heart rhythm despite beta blockade
  * Creatinine >1.6 mg/dl
  * Allergy to iodinated contrast medium
  * Inability to lie flat

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with suspected or known myocardial ischemia
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-09; Primary Completion 2017-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy measures of cardiac CT perfusion techniques | 1 month
  Diagnostic performance includes sensitivity, specificity, positive and negative predictive values, and receiver operator curve area under the curve [ROC AUC]. The highest ROC AUC will be considered the best diagnostic performance and will be compared statisically using the c-statistic.

SECONDARY OUTCOMES:
Minimal number of images needed for CT perfusion | 1 month
  Using modeling techniques, we will determine the least number of images needed for each CT perfusion technique to maintain diagnostic accuracy. The fewer number of images will correspond to a lower radiation dose.
Diagnostic accuracy of CCTA and CT perfusion compared to PET perfusion imaging alone | 1 month
  Incremental diagnostic accuracy changes with CCTA + CT perfusion compared to PET perfusion alone.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States